CLINICAL TRIAL: NCT06756347
Title: Comparative Analysis of Ultrasound-Guided Versus Landmark-Based Techniques for Regional Anesthesia in Egyptian Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tarek Ashraf Ibrahim Abd Al-Hafiz, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: US-Guided vs Land mark RA
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Group (Active Comparator): Patients receiving ultrasound-guided brachial plexus blocks .o Procedure performed using a high-frequency linear ultrasound probe.Real-time visualization of the brachial plexus for precise anesthetic delivery
  Interventions: Procedure: Patients receiving landmark-based brachial plexus blocks; Drug: Bupivacaine
- Landmark-Based Group (Active Comparator): Patients receiving landmark-based brachial plexus blocks.o Procedure performed based on anatomical landmarks and palpation, without imaging assistance
  Interventions: Procedure: Landmark-Based Brachial Plexus Block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Patients receiving landmark-based brachial plexus blocks — The operator will visualize anatomical structures in real time, identify the brachial plexus (supraclavicular approach), and guide the needle to the injection site under direct ultrasound visualization
  Arms: Ultrasound-Guided Group
Procedure: Landmark-Based Brachial Plexus Block — The operator will identify anatomical landmarks (e.g., interscalene groove, supraclavicular fossa) using palpation and surface anatomy. The needle will be inserted based on these landmarks, with no direct visualization of internal structures.
  Arms: Landmark-Based Group
Drug: Bupivacaine — injected in both group as local anesthetic agent ( at a standardized concentration and volume) to ensure comparability.

SUMMARY:
Regional anesthesia is a cornerstone in modern surgical practices due to its ability to provide effective pain management and reduce reliance on general anesthesia. Traditional landmark-based techniques, widely used due to their simplicity and cost-effectiveness, rely on surface anatomy and palpation to guide needle placement. However, these techniques are associated with a higher risk of complications, including failed blocks and nerve injuries.

Ultrasound-guided techniques have emerged as a safer, more precise alternative, offering real-time visualization of anatomical structures. Studies suggest that ultrasound guidance improves the success rate, reduces procedural time, and minimizes complications. Despite global advancements in ultrasound-guided regional anesthesia, limited research addresses its efficacy and safety specifically in Egyptian patients, whose unique anatomical and physiological characteristics may influence outcomes.

This study seeks to fill this knowledge gap and provide evidence-based guidance tailored to this population, focusing on brachial plexus blocks.

DETAILED DESCRIPTION:
Regional anesthesia is a cornerstone in modern surgical practices due to its ability to provide effective pain management and reduce reliance on general anesthesia. Traditional landmark-based techniques, widely used due to their simplicity and cost-effectiveness, rely on surface anatomy and palpation to guide needle placement. However, these techniques are associated with a higher risk of complications, including failed blocks and nerve injuries.

Ultrasound-guided techniques have emerged as a safer, more precise alternative, offering real-time visualization of anatomical structures. Studies suggest that ultrasound guidance improves the success rate, reduces procedural time, and minimizes complications. Despite global advancements in ultrasound-guided regional anesthesia, limited research addresses its efficacy and safety specifically in Egyptian patients, whose unique anatomical and physiological characteristics may influence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ● Adult patients aged 18-65 years undergoing upper limb surgery requiring brachial plexus block.

  * Patients capable of providing informed consent

Exclusion Criteria:

* ● Patients with contraindications to regional anesthesia (e.g., infection at the site, severe coagulopathy).

  * History of severe allergic reactions to local anesthetics.
  * Anatomical abnormalities affecting the brachial plexus block.
  * Obesity (BMI > 35) or other conditions that might confound results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 30 minutes
  Proportion of patients achieving adequate anesthesia (complete sensory block) within 30 minutes of administration.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sivashanmugam T, Ray S, Ravishankar M, Jaya V, Selvam E, Karmakar MK. Randomized Comparison of Extrafascial Versus Subfascial Injection of Local Anesthetic During Ultrasound-Guided Supraclavicular Brachial Plexus Block. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):337-43. doi: 10.1097/AAP.0000000000000264. PMID 26066385